CLINICAL TRIAL: NCT00894608
Title: Letrozole Combined With Gn for Ovarian Hyperstimulation Undergoing IVF/ICSI in Patients With PCOS
Brief Title: Letrozole Combined With Gonadotropins (Gn) for Ovarian Stimulation Undergoing in Vitro Fertilization/Intracytoplasmic Sperm Injection (IVF/ICSI) in Patients With Polycystic Ovary Syndrome (PCOS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Yunyang Medical College (Other)
Responsible Party: reproductive medicine research center, renmin hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: a00949200
Record Dates: First submitted 2009-05-05; First posted 2009-05-07 (Estimated); Last update posted 2009-05-07 (Estimated); Status verified 2009-05

CONDITIONS: Polycystic Ovarian Syndrome
Keywords: letrozole; ovarian stimulation; PCOS; IVF-ET
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Letrozole; Gonadotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- letrozole protocol (Experimental): patients in letrozole protocol for ovarian stimulation with letrozole combined with gonadotropins
  Interventions: Drug: letrozole + gonadotropins
- long GnRHa protocol (Experimental): patients in long GnRHa protocol for ovarian stimulation with Gnrha and gonadotropins
  Interventions: Drug: GnRHa + gonadotropins

INTERVENTIONS:
Drug: letrozole + gonadotropins — patients in letrozole protocol for ovarian stimulation with letrozole combined with gonadotropins
  Arms: letrozole protocol
Drug: GnRHa + gonadotropins — patients in long GnRHa protocol for ovarian stimulation with GnRHa and gonadotropins
  Arms: long GnRHa protocol

SUMMARY:
The purpose of this study is to determine whether letrozole combined with gonadotropins are effective in the ovarian hyperstimulating for IVF/ICSI in patients with PCOS.

DETAILED DESCRIPTION:
Polycystic ovarian syndrome (PCOS) occurs in 4% to 7% of all women of reproductive age and 20% of women presenting with anovulatory infertility. A significant proportion of these women will ultimately need assisted reproductive techniques. Various protocols of ovarian stimulation such as step up protocol, coasting, GnRH antagonists et al have been proposed for optimizing IVF results in patients with PCOS. The results of these studies have shown it not to be satisfied. The preliminary studies have proven that Letrozole, a potent and highly specific nonsteroidal aromatase inhibitor, could successfully induce ovulation in women with polycystic ovary syndrome. In spite of only a little study research of letrozole in IVF/ICSI cycle, for poor ovarian responders, addition of letrozole improved ovarian response to FSH and reduced gonadotrophin dose required for COH without having a negative impact on pregnancy rates. These reports prompted us to hypothesize that adjunctive use of letrozole in COH protocol for patients with PCOS would minimize the gonadotrophin dose, and consequently the cost, and lower the risk of OHSS in a IVF/ICSI treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

* patients with PCOS

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Cycle cancellation rate, number of oocytes retrieved, fertilization rate, embryo quality, clinical pregnancy, implantation rates and OHSS rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: zhang changjun, doctor, Study Director — renmin hospital,yunyang medical college
Locations (1):
- Reproductive Medcine Research Center, Shiyan, Hubei, China